CLINICAL TRIAL: NCT03179410
Title: PD-L1 Inhibition as ChecKpoint Immunotherapy for NeuroEndocrine Phenotype Prostate Cancer
Acronym: PICK-NEPC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andrew J. Armstrong, MD (Other)
Responsible Party: Sponsor-Investigator, Andrew J. Armstrong, MD, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00080869
Record Dates: First submitted 2017-06-05; First posted 2017-06-07 (Actual); Results first posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-02

CONDITIONS: Prostate Cancer
Keywords: metastatic castrate-resistant prostate cancer (mCRPC); neuroendocrine prostate cancer (NEPC)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Neuroendocrine prostate cancer (NEPC) (Experimental): Subjects with neuroendocrine prostate cancer (NEPC). Avelumab will be administered intravenously at a dose of 10 mg/kg every 2 weeks.
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — 10 mg/kg intravenously every 2 weeks

SUMMARY:
The purpose of this study is to assess the safety and efficacy of avelumab in patients with metastatic neuroendocrine-like prostate cancer. Eligible men will be started on avelumab every 2 weeks and will stay on therapy until progression or intolerable side effects. The central hypothesis is that PD-L1 inhibition with avelumab will be efficacious based on radiographic responses in a subset of men with metastatic neuroendocrine-like prostate cancer and be reasonably well tolerated, meeting criteria for further study in larger phase 2 and 3 trials based on meeting pre-specified efficacy rates and prolonged PFS in some men.

ELIGIBILITY:
Inclusion Criteria:

1. Neuroendocrine-like prostate cancer, based on histology OR based on clinical presentation as defined by meeting one of the two below criteria. All subjects must submit their primary tumor or metastatic biopsy pathology specimens to the Duke Cancer Institute where they will be centrally reviewed by Duke Pathology. Central Duke pathologic review is not required for screening but rather for confirmation of histologic subtype. Local pathologic review is sufficient for eligibility determination.

   1. Criterion 1: Presence of 1 of 3 histologically proven diagnoses: 1) Primary small cell carcinoma of the prostate, defined by classic histologic features such as small tumor cells with scanty cytoplasm, darkly stained nuclei with homogeneous chromatin pattern. The tumor cells do not form glandular structure but grow as solid sheets with frequent mitotic figures and necrosis; 2) Intermediate atypical carcinoma of the prostate, which has histologic features distinct from small cell carcinoma or adenocarcinoma. The tumor grows as solid sheets or vague glandular structures. The tumor cells have moderate amounts of cytoplasm and centrally located, round and regular nuclei with fine, granular and homogeneous chromatin. Mitosis and necrosis are absent; 3) mixed histology tumors of the prostate, containing both adenocarcinoma and neuroendocrine or small cell components.
   2. Criterion 2: Presence of histologically proven adenocarcinoma of the prostate without any sign of neuroendocrine or small cell histology that is radiographically progressing despite castrate levels of testosterone (<50 ng/mL) with the following poor risk features:

   i. Prior progression despite therapy with either abiraterone acetate and/or enzalutamide ii. At least one of the following: 1) Liver metastases; 2) Bulky radiographic progression (≥2 cm short axis lymph nodes or ≥1 cm long axis visceral metastases) combined with low serum PSA (<10ng/mL); 3) High serum LDH (>1X upper limit of normal).
2. Measurable disease as defined by modified PCWG3 using iRECIST criteria
3. Available tumor tissue for pathologic review and correlative studies. Tumor tissue (localized or metastatic) does not need to be received but rather identified and available (slides and/or blocks) to be sent to Duke.
4. Documented progressive metastatic CRPC based on at least one of the following criteria:

   1. PSA progression defined as 25% increase over baseline value with an increase in the absolute value of at least 2.0 ng/mL that is confirmed by another PSA level with a minimum of a 1 week interval and a minimum PSA of 2.0 ng/mL. Note: If confirmed rise is the only indication of progression, a minimal starting value of 1.0 ng/mL is acceptable, unless pure small-cell carcinoma.
   2. Soft-tissue progression based on new lesions or growth of existing soft tissue metastases.
   3. Progression of bone disease (evaluable disease) or (new bone lesion(s)) by bone scan.
5. Castrate levels of serum total testosterone (<50 ng/dl) OR ongoing documented ADT unless pure small cell prostate cancer is present.
6. Previous use of radiation to metastatic site(s) at any time prior to enrollment is allowed, provided that this site is not the only measurable disease present or unless that solitary site is progressing following radiation.
7. Patients should have received at least one line of approved chemotherapy and/or hormonal therapy
8. Previous cytotoxic chemotherapy including cisplatin, carboplatin, oxaliplatin, etoposide, docetaxel, cabazitaxel, and gemcitabine is allowed, up to 3 prior regimens.
9. Karnofsky performance status of 70 or higher.
10. Acceptable initial laboratory values within 14 days of Cycle 1 Day 1 according to the below table:

    ANC ≥ 1500/µl Hemoglobin ≥ 9.0 g/dL(prior transfusion permitted) Platelet count ≥ 100,000/µl Creatinine ≤ 2.0 x the institutional upper limit of normal (ULN) OR creatinine clearance >30 ml/min Potassium ≥ 3.5 mmol/L (within institutional normal range) Bilirubin ≤ 1.5 x ULN (unless documented Gilbert's disease) SGOT (AST) ≤ 2.5x ULN, or <5x ULN in patients with documented liver metastases SGPT (ALT) ≤ 2.5x ULN or <5x ULN in patients with documented liver metastases
11. Age >18
12. Highly effective contraception for male subjects with childbearing potential throughout the study and for at least 60 days after last avelumab treatment administration if the risk of conception exists.
13. Willing and able to provide written informed consent and HIPAA authorization for the release of personal health information.
14. Life expectancy of over 3 months as determined by treating physician.

Exclusion Criteria:

1. Prior usage of PD-1 inhibitors, programed-death ligand 1 and/or 2 inhibitors, CTLA-4 inhibitors including but not limited to ipilimumab, nivolumab, avelumab, durvalumab, tremelimumab, and pembrolizumab.
2. Active on-going immunologic or autoimmune disease including but not limited to systemic or cutaneous lupus erythematosus, cutaneous psoriasis, psoriatic arthritis, rheumatoid arthritis, scleroderma, sicca syndrome, polymyalgia rheumatica, polyarteritis nodosa, granulomatous polyangiitis, microscopic polyangiitis, polyarteritis nodosa, temporal arteritis, giant cell arteritis, dermatomyositis, Kawasaki disease.
3. Previous malignancy within 3 years other than non-melanomatous skin cancers or cancers of low malignant potential such as non-invasive urothelial carcinoma.
4. Any other on-going chemotherapeutic, biologic, radiopharmaceutical, or investigational agent currently or within 28 days of Cycle 1 Day 1.
5. Prior use of abiraterone and other hormonal agents used to treat prostate cancer are permitted but abiraterone acetate should be stopped prior to study treatment initiation.
6. Current usage of immunosuppressant medication except for a) intranasal, inhaled, and topical corticosteroids and b) systemic corticosteroids equivalent to ≤ 10 mg/day of prednisone, c) steroids as premedication for hypersensitivity reactions (e.g. CT scan premedication).
7. Prior organ transplantation including allogeneic stem-cell transplants.
8. Active bacterial or viral infections requiring systemic therapy.
9. Current active infections with HIV/AIDS, Hepatitis B, and Hepatitis C requiring treatment.
10. Live virus vaccination within 4 weeks of the first dose of avelumab (inactivated vaccines are allowed).
11. Known prior hypersensitivity to the investigational product or any component formulations, including known severe hypersensitivity reactions to monoclonal antibodies.
12. Clinically significant (i.e. active) cardiovascular disease: cerebral vascular accident (<6 months prior to enrollment), myocardial infarction (<6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
13. Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, Grade 2 anemia, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.
14. Other severe acute or chronic medical conditions including colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Armstrong, MD, ScM, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Brown LC, Halabi S, Somarelli JA, Humeniuk M, Wu Y, Oyekunle T, Howard L, Huang J, Anand M, Davies C, Patel P, Staats J, Weinhold KJ, Harrison MR, Zhang T, George DJ, Armstrong AJ. A phase 2 trial of avelumab in men with aggressive-variant or neuroendocrine prostate cancer. Prostate Cancer Prostatic Dis. 2022 Apr;25(4):762-769. doi: 10.1038/s41391-022-00524-7. Epub 2022 Mar 15. PMID 35292724

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm-arm Phase II Study of Avelumab: Subjects with metastatic neuroendocrine-like prostate cancer will be treated with Avelumab intravenously at a dose of 10 mg/kg every 2 weeks.
Period: Overall Study
Arm/Group | Single Arm-arm Phase II Study of Avelumab
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm-arm Phase II Study of Avelumab
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 71 [51 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Prior PSA [Median (Full Range); unit: ng/ml] | 53.6 [0.0 to 393.0]
Karnofsky Performance Status Score [Median (Full Range); unit: units on a scale] — Karnofsky score for performance (KPS) status calculator scale runs from 100 to 0 where 100 means the patient's condition is normal and 0 indicates death. Higher the score, better is the condition.
  units on a scale | 90 [80 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Response as Determined by iRECIST
Description: Overall response rate is determined by radiographic response assessment utilizing modified Prostate Cancer Working Group 3 (PCWG3) using Immune Response Evaluation Criteria In Solid Tumors Criteria (iRECIST 1.1). iRECIST is the modified RECIST 1.1 for immune-based therapeutics, to measure radiographic response rate in men with metastatic prostate cancer. Patients alive who had not progressed as of the last follow-up, had PFS censored at the last follow-up date. There are five categories overall responses:
  iCR: immune complete response achieved with disappearance of all target lesions iCPD: immune confirmed progressive disease when there is either 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions iSD: immune stable disease in the absence of CR or PD iUPD: immune unconfirmed progressive disease when PD is unconfirmed NE: not evaluable
Time Frame: baseline to end of treatment (approximately 6 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm-arm Phase II Study of Avelumab
Number analyzed (Participants) | 15
Participants
  iCR: immune complete response | 1
  iCPD: immune confirmed progressive disease | 1
  iSD: immune stable disease | 3
  iUPD: immune unconfirmed progressive disease | 9
  NE: not evaluable | 1

2. Secondary Outcome: Efficacy of PD-L1 Inhibition With Avelumab as Determined by RECIST1.1
Description: Overall response rate is determined by radiographic response assessment utilizing Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1). Patients alive who had not progressed as of the last follow-up, had PFS censored at the last follow-up date. There are four overall response categories:
  Complete Response (CR): disappearance of all target and non-target lesions Progressive Disease (PD): 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions Stable Disease (SD): In the absence of CR and PD Unevaluable (NE)
Time Frame: baseline to end of treatment (approximately 6 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm-arm Phase II Study of Avelumab
Number analyzed (Participants) | 15
Participants
  Complete Response (CR) | 1
  Progressive Disease (PD) | 10
  Stable Disease (SD) | 3
  Unevaluable (NE) | 1

3. Secondary Outcome: Radiographic Progression Free Survival (rPFS)
Description: Radiographic progression free survival (rPFS) as determined by PCWG3 and RECISTS1.1 criteria. Radiographic progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Patients alive who had not progressed as of the last follow-up had PFS censored at the last follow-up date. Median rPFS was estimated using a Kaplan-Meier curve.
Time Frame: baseline to end of treatment (approximately 6 months)
Measure: Median (Full Range); unit: month
Arm/Group | Single Arm-arm Phase II Study of Avelumab
Number analyzed (Participants) | 15
month | 1.8 [1.6 to 2.0]

4. Secondary Outcome: Overall Survival
Description: Length of patient's life after starting study
Time Frame: Up to 23.5 months
Measure: Median (Full Range); unit: month
Arm/Group | Single Arm-arm Phase II Study of Avelumab
Number analyzed (Participants) | 15
month | 7.4 [2.8 to 12.5]

5. Secondary Outcome: Toxicity and Safety of PD-L1 Inhibition With Avelumab in Men With Metastatic Neuroendocrine-like Prostate Cancer
Description: Number of Participants with Adverse Events
Time Frame: 28 days post-treatment (approximately 7 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm-arm Phase II Study of Avelumab
Number analyzed (Participants) | 15
Participants | 15

ADVERSE EVENTS:
Time Frame: Up to 30 days post last day of dosing
Arm/Group | Single Arm-arm Phase II Study of Avelumab
All-Cause Mortality (participants affected / at risk) | 9/15
Serious Adverse Events (participants affected / at risk) | 9/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm-arm Phase II Study of Avelumab (N=15)
Hypocalcemia (Metabolism and nutrition disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Delirium (Psychiatric disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Anemia (Blood and lymphatic system disorders) | 2
Fever (General disorders) | 2
Surgical and medical procedures - Other Specify; Brain mass removal (Surgical and medical procedures) | 1
Glucose intolerance (Metabolism and nutrition disorders) | 1
Neoplasms benign malignant and unspecified (incl cysts and polyps) - Other Specify; Brain mets (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thromboembolic event (Vascular disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Syncope (Nervous system disorders) | 1
Pericarditis (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm-arm Phase II Study of Avelumab (N=15)
Anemia (Blood and lymphatic system disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Blurred vision (Eye disorders) | 1
Eye disorders - Other, Specify: DIPLOPIA (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Bloating (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other, Specify: TOOTH FRACTURE (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 3
Chills (General disorders) | 3
Fatigue (General disorders) | 6
Fever (General disorders) | 2
Infusion related reaction (General disorders) | 9
Localized edema (General disorders) | 2
Malaise (General disorders) | 1
Pain (General disorders) | 1
Infections and infestations - Other, Specify: C. DIF (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 4
Fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 3
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 1
Creatinine increased (Investigations) | 3
Investigations - Other, Specify: POSITIVE FOR BLOOD IN STOOL (Investigations) | 1
Weight loss (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 1
Glucose intolerance (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal and connective tissue disorder - Other, Specify: GROIN STRAIN (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, Specify: MUSCLE CRAMPS (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 2
Encephalopathy (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Nervous system disorders - Other, Specify: CAUDA EQUINA (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 1
Urine discoloration (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, Specify: YAWNING (Respiratory, thoracic and mediastinal disorders) | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, Specify: ABRASION RIGHT ELBOW (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, Specify: LEFT NOSTRIL SCAB (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, Specify: MONS PUBIS (HERPES) (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, Specify: RASH LEFT KNEE, MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, Specify: WOUND ON BACK (Skin and subcutaneous tissue disorders) | 1
Surgical and medical procedures - Other, Specify: RIGHT PERCUTANEOUS NEPHROSTOMY TUBE PLACED (Surgical and medical procedures) | 1
Flushing (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/10/NCT03179410/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/10/NCT03179410/Prot_SAP_001.pdf